CLINICAL TRIAL: NCT06311344
Title: Filling Key Research Gaps With Clinical Implications in Mansonellosis and Schistosomiasis: a Network Approach
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-06
Record Dates: First submitted 2024-03-06; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Schistosoma Mansoni
MeSH Terms: conditions — Schistosomiasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological samples (Other): M. perstans microfilariae and Schistosoma spp eggs, obtained from the routine diagnostic procedures carried out on patients, specifically migrants and travellers, visited in the centres participating to this study
  Interventions: Diagnostic Test: Molecular biology analyses

INTERVENTIONS:
Diagnostic Test: Molecular biology analyses — Samples of M. perstans microfilariae will be processed by PCR to investigate the presence (or absence) of Wolbachia using a set of primers targeting the genes ftsZ and 16S and optimized using reference material during the first year of the study. Samples of Schistosoma eggs from urine and feces will be processed for DNA extraction. Each sample will be genetically characterised by multi locus analysis of the mitochondrial cox1 region and the nuclear ITS and 18S rRNA regions. PCR products will be analysed by agarose gel electrophoresis and selected amplicons will be purified and Sanger sequenced. For the individuation of Schistosoma hybrids, the nuclear DNA for each sample will be confirmed by analysis of the species-specific polymorphic positions of the ITS1+2 and 18S. The mitochondrial and nuclear DNA genetic profiles for each individual sample will be recorded to determine the species involved in the infections and also any hybrid schistosomes

SUMMARY:
This is an experimental, multicenter, non-profit study promoted by the Department of Infectious and Tropical Diseases of the IRCCS (Istituto di Ricerca e Cura a carattere scientifico) Sacro Cuore Don Calabria of Negrar which aims to evaluate the presence of endosymbiont Wolbachia in circulating microfilariae obtained from biological samples of individuals infected with M .perstans and the presence of infection with hybrid Schistosoma species in the population of Schistosoma eggs isolated from biological samples of patients with active schistosomiasis.

ELIGIBILITY:
Inclusion criteria:

* samples from patients who gave consent to the storage and use for research purposes of their samples. In the case a network centre necessitates a template for the storage and use for research purposes of their samples;
* samples collected before any treatment with praziquantel and/or benzimidazole and/or avermectin and/or diethylcarbamazine and/or doxycycline drug;
* samples collected and stored in conditions suitable for this study (Annex 2);
* known country of birth of the patient or of most likely infection (if different from the country of birth)

Exclusion criteria:

- no compliance with at least one of the above-mentioned inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of M. perstans microfilariae | Baseline
  Number of samples, defined as the whole M. perstans microfilariae retrieved from one blood sample from each patient, positive for the presence of Wolbachia as assessed by PCR.
Percentage of M. perstans microfilariae | Baseline
  Percentage of samples, defined as the whole M. perstans microfilariae retrieved from one blood sample from each patient, positive for the presence of Wolbachia as assessed by PCR.
Number of Schistosoma eggs | Baseline
  Number of samples defined as the whole Schistosoma eggs retrieved from one stool or urine sample from each patient, positive for the presence Schistosoma hybrid species.
Percentage of Schistosoma eggs | Baseline
  Percentage of samples defined as the whole Schistosoma eggs retrieved from one stool or urine sample from each patient, positive for the presence Schistosoma hybrid species.

SECONDARY OUTCOMES:
Number of samples positive for Wolbachia | Baseline
  number of samples, defined as the whole M. perstans microfilariae retrieved from one blood sample from each patient, positive for the presence of Wolbachia as assessed by PCR, by country of origin of the patient or most likely country of infection.
Percentage of samples positive for Wolbachia | Baseline
  Percentage of samples, defined as the whole M. perstans microfilariae retrieved from one blood sample from each patient, positive for the presence of Wolbachia as assessed by PCR, by country of origin of the patient or most likely country of infection.
Number of samples positive for Schistosoma hybrid species | Baseline
  number of samples defined as the whole Schistosoma eggs retrieved from one stool or urine sample from each patient, positive for the presence Schistosoma hybrid species by country of origin of the patient or most likely country of infection.
Percentage of samples positive for Schistosoma hybrid species | Baseline
  percentage of samples defined as the whole Schistosoma eggs retrieved from one stool or urine sample from each patient, positive for the presence Schistosoma hybrid species by country of origin of the patient or most likely country of infection.
Identification of hybrid species of Schistosoma spp. | Baseline
  Identification of hybrid species from each parental species of Schistosoma spp.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Sacro Cuore Don Calabria hospital, Negrar, Verona, Italy